CLINICAL TRIAL: NCT04808856
Title: Treatment of Refractory Gout With Adrenocorticotropic Hormone or Methylprednisolone
Brief Title: Treatment of Refractory Gout With ACTH or Methylprednisolone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTH
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Adrenocorticotropic Hormone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTH (Experimental): Adrenocorticotropic Hormone
  Interventions: Drug: Adrenocorticotropic Hormone
- Methylprednisolone (Active Comparator): Methylprednisolone
  Interventions: Drug: Methylprednisolone Injection

INTERVENTIONS:
Drug: Adrenocorticotropic Hormone — Adrenocorticotropic Hormone Injection 25u qd iv *3d
  Arms: ACTH
Drug: Methylprednisolone Injection — Methylprednisolone Injection 40mg qd iv *3d
  Arms: Methylprednisolone

SUMMARY:
To clarify the therapeutic effect and safety evaluation of ACTH in refractory gouty arthritis and special population, and to explore its mechanism of action.

DETAILED DESCRIPTION:
When patients with acute gout have multiple comorbidities and complications , traditional treatment methods are often contraindicated . From the current clinical research evidence , we have seen the non-inferior effect of ACTH on glucocorticoids and non-steroidal anti-inflammatory drugs in the treatment of acute gout , as well as the good safety and extensive anti-inflammatory effect in addition to efficacy . Therefore , we designed this study to update and improve the treatment of acute gout attacks , and to try to clarify the mechanism of action .

ELIGIBILITY:
Inclusion Criteria:

* (123 items and 1 item from 4-7 are met simultaneously) :

  1. Meet the 2015 ACR/EULAR classification diagnostic criteria for gout
  2. Acute gouty arthritis
  3. Age ≥18
  4. Repeated attacks and prolonged pain (more than 1 month);
  5. poor response or intolerance to colchicine or NSAIDs;
  6. Liver and kidney dysfunction;
  7. Old age;

Exclusion Criteria:

* 1) History of gastrointestinal bleeding and active ulcer 2) The application history of glucocorticoids and ACTH in 1 month before screening 3) Pregnancy and lactation 4) Drug and alcohol abuse 5) Malignant tumor (treated or untreated within 5 years) 6) Mental illness inability to communicate or have language barriers and inability to fully understand and cooperate 7) negligent compensatory heart failure, unstable angina pectoris, stroke, transient ischemic attack, myocardial infarction, and severe arrhythmia occurred within 6 months 8) The investigator did not consider it appropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of pain | 7 days
  Visual analogue scale (VAS 0-10)
Arthritis score | 7 days
  Arthritis (redness and swelling fever 0-3) score

SECONDARY OUTCOMES:
Recurrence rate | 1 month
  Recurrence rate (3d, 7d, 2w, 1m follow-up; recurrence within 1m was defined as recurrence)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, M.D Ph.D, Principal Investigator — Shanghai Tenth People' Hospital
Locations (1):
- Shanghai Tenth People's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No